CLINICAL TRIAL: NCT05386745
Title: A Feasibility Study Evaluating an Online Physical Activity Intervention for Young Adults With Low Mood and/or Depression Engaged in Community Primary Clinical Care
Brief Title: Feasibility Study of an Online Physical Activity Intervention for Youth With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0301
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-11

CONDITIONS: Low Mood; Mild Depression; Moderate Depression; Inactivity, Physical
MeSH Terms: conditions — Consciousness Disorders; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An online, asynchronous, self-paced, 10-week long, physical activity intervention.
  Interventions: Behavioral: physical activity
- Control (No Intervention): A waitlist control; continue with life/activity as usual. Control participants will receive access to the intervention at 10 weeks following all measurements.

INTERVENTIONS:
Behavioral: physical activity — A series of 10 weekly psychoeducational modules including information on psychosocial determinants of physical activity engagement, adherence and maintenance, as well as a number of other behaviour change tools, like reflection activities.
  Arms: Intervention

SUMMARY:
Physical activity (PA) has recently been established as both a primary intervention for mild to moderate, and a secondary therapy for moderate to severe Major Depressive Disorder (MDD; Fortier et al., 2020). Those with mental health disorders do not on average achieve recommended levels of PA (Hallgren et al., 2016), and exercise prescription is extremely lacking in clinical care (Stanton, Reaburn, & Happell, 2015; Stanton et al., 2018). Theory-based behavioural interventions have proven to be an effective tool for improving physical activity levels in clinical populations (Glowacki, et al., 2017; Stanton et al., 2015). More research is needed to understand PA intervention effectiveness for MDD patients (Glowacki et al., 2017), support integration of such behavioural treatments with primary care (Lederman et al., 2017), and address growing concerns regarding mental health during the global pandemic and beyond (Boyce, 2021). This community-based study examines the feasibility of a co-designed, 10-week, asynchronous, web-based beta platform PA intervention for patients with experience of low mood and/or mild to moderate depression, and will provide important parameters for a future randomized-controlled trial (RCT). Primary outcome measures will focus on acceptability and feasibility, including recruitment and retention rates. Secondary measures will include physical activity and depression symptom severity. Behavioural predictors of PA are to be evaluated as tertiary outcomes. Questionnaires will include an adapted participant experience measure, Godin Leisure-Time Exercise Questionnaire, and the Patient Health Questionnaire-9. This study features a controlled baseline, post-intervention evaluative design with an embedded quantitative process evaluation with a waitlist control. Participants will be young adults with experience of low mood and/or mild to moderate depression, 19-30 years of age, with access to a device with internet, English speaking, living within British Columbia, CAN., and falling below the minimum Canadian recommendations for PA. Study recruitment will primarily be facilitated by multiple youth mental health primary and community care clinics. This study will contribute to understanding of acceptable, efficacious, behaviour-based and mobile health intervention approaches for young adults with depression. It will also provide young people with a platform to share invaluable feedback to direct innovations in their own alternative care and mental health treatment. If outcome benchmarks set based on previous literature are met or exceeded for each of recruitment, retention, and acceptability, and depressive symptoms trend downwards for intervention participants, then a future randomized controlled trial exploring principally mental health outcomes will be recommended.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 19-30 years
* experience of low mood and/or mild to moderate depression (no diagnosis required)
* report falling below minimum Canadian public health recommendations for PA consistently over the past 6 months
* report no contraindications to physical activity (based on the completion of the Physical Activity Readiness Questionnaire administered at screening)
* do not report any manic or psychotic episodes within the past 6 months
* do not report any substance or alcohol abuse within the past 6 months
* have access to a device with an internet connection
* reside in British Columbia currently
* fluent in English

Exclusion Criteria:

* be young adults, 19-30 years of age,
* currently reside in British Columbia,
* self-identify as someone with experience of depression (ranging from low mood and/or depressive symptoms to a formal mild to moderate Major Depressive Disorder diagnosis according to the Diagnostic and Statistical Manual of Mental Health Disorders-V)
* report no manic episode(s) or psychosis in the past 6 months,
* fall below the minimum Canadian public health recommendations for PA (Ross et al., 2020) for at least six months prior to screening,
* have access to a device with internet access, AND
* English speaking.

No exclusion criteria for sex, gender, medications, race or religion will be applied. There will be no contraindications to PA after screening with the Physical Activity Readiness Questionnaire (PAR-Q).

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 10 weeks
  outcome related to trial feasibility
Retention Rate | 10 weeks
  outcome related to trial feasibility
Experience Measure | 10 weeks
  outcome related to trial acceptability

SECONDARY OUTCOMES:
Depression Severity | 10 weeks
  measured with the Patient Health Questionnaire-9 (min.=0, max.=27, lower scores indicate fewer symptoms of depression)
Physical Activity Levels | 10 weeks
  measured with the Godin Leisure Time Exercise Questionnaire (min.=0, max.=N/A, higher scores indicate increased physical activity)

OTHER OUTCOMES:
Psychosocial Factors Predicting Physical Activity Behaviour | 10 weeks
  measured with the Multi-Process Action Control Framework which included various constructs and measurements scales, e.g., affective and instrumental attitude (min.=1, max.=7, higher scores indicate increased positively-valenced attitude; Ajzen 2002; Rhodes and Courneya 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Aleah B Ross, BSc, Study Director — University of Victoria; Ryan E Rhodes, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No